CLINICAL TRIAL: NCT00382512
Title: A Randomized, Placebo-Controlled, Single-Blind, Parallel-Group Study to Evaluate the Effects of 12 Weekly Subcutaneous Doses of 1.0 mg/kg Efalizumab on Immune Responses in Subjects With Moderate Plaque Psoriasis
Brief Title: A Study to Evaluate the Effects of Efalizumab on Immune Responses in Subjects With Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACD2244g
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2006-09-29 (Estimated); Status verified 2006-09

CONDITIONS: Plaque Psoriasis
Keywords: Moderate Plaque Psoriasis
MeSH Terms: interventions — efalizumab

INTERVENTIONS:
Drug: Raptiva (efalizumab)

SUMMARY:
This is a Phase I, randomized, placebo-controlled, single blind, parallel group, single-center study designed to evaluate immune responses during and after administration of 12 weekly SC doses of 1.0 mg/kg efalizumab in subjects with moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Plaque psoriasis covering 8%-15% of the total BSA
* Diagnosis of plaque psoriasis for at least 6 months
* Body weight of ≤140 kg
* 18 to 65 years old
* For women of childbearing potential and men who may father children, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study (the following methods of contraception are acceptable: condom; abstinence; oral, implantable or injectable contraceptives by the sexual partner; IUD, female condom, diaphragm with spermicide, cervical cap; a sterile sexual partner)
* Willingness to hold sun exposure reasonably constant and to avoid use of tanning booths or other UV light sources during the study
* History of tetanus vaccination

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* History of severe allergic or anaphylactic reactions to humanized monoclonal antibodies or fusion proteins that contain an Ig Fc region
* Clinically significant psoriasis exacerbation during screening or at the time of enrollment
* History of or ongoing uncontrolled bacterial, viral, fungal, or atypical mycobacterial infection
* History of opportunistic infections (e.g., systemic fungal infections, parasites)
* Seropositivity for human immunodeficiency virus (HIV)
* Pregnancy or lactation
* White blood cell (WBC) count <4000/uL or >14,000/uL
* Seropositivity for hepatitis B or C virus
* Hepatic enzymes ≥3 times the upper limit of normal
* Tetanus or pneumococcal vaccination during the 6 months prior to the start of the study (Treatment Day 0) or failure to complete a primary series of tetanus immunizations
* Known hypersensitivity reaction to tetanus or diphtheria toxoid
* Known hypersensitivity to any of the administered vaccinations or their components
* History of active tuberculosis (TB) or currently undergoing treatment for TB
* Positive purified protein derivative (PPD) (tuberculin) testing at screening (as defined by CDC Guidelines, see Appendix C for test assessment criteria and listing of high-risk groups)
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders
* Treatment with efalizumab (anti-CD11a) within the last 12 months
* Previous administration of <phi>X174
* Diagnosis of hepatic cirrhosis, regardless of cause or severity
* Serum creatinine ≥2 times the upper limit of normal
* Hospital admission for cardiac disease, stroke, or pulmonary disease within the last year
* History of substance abuse within the last 5 years as judged by the Principal Investigator
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug
* Systemic therapy for psoriasis (Screening Day -28 through FU Day 98)
* Systemic immunosuppressive drugs for any indications (Screening Day -28 through FU Day 98)
* Live virus or bacteria vaccines other than protocol specified (Screening Day -14 through Treatment Day 84)
* Other vaccines or allergy desensitization (must be scheduled at least 14 days prior to Treatment Day 0 or after FU Day 98)
* Other experimental drugs or treatments (within 90 days or five half-lives, whichever is longer, prior to Treatment Day 0 and through FU Day 98)
* <beta>-Blockers, angiotensin-converting enzyme (ACE) inhibitors, quinidine, antimalarial drugs, or lithium (if clinically indicated, such medications are allowed but the dosage should be held constant between Screening Day -28 and Treatment Day 84)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-05

PRIMARY OUTCOMES:
Mean concentrations of anti-<phi>X174 antibodies in the FU period 2 weeks after the FU Day 70 vaccinations in Group A compared with mean antibody concentrations 2 weeks after the Treatment Day 63 vaccination in Group C
Mean concentrations of anti-<phi>X174 antibodies in the FU period 2 weeks after the FU Day 70 vaccination in Group B compared with mean antibody concentrations 2 weeks after the Treatment Day 63 vaccination in Group C.

SECONDARY OUTCOMES:
Characterization of mean concentrations of anti-<phi>X174 antibodies 2 weeks after the FU Day 42 vaccination in Group A compared with mean antibody concentrations 2 weeks after the Treatment Day 35 vaccination in Group C
Characterization of mean concentrations of anti-<phi>X174 antibodies 2 weeks after the FU Day 42 vaccination in Group B compared with mean antibody concentrations 2 weeks after the Treatment Day 35 vaccination in Group C
Characterization of mean anti-<phi>X174 concentrations 2 and 4 weeks after the first and 2 and 4 weeks after the second <phi>X174 vaccinations during efalizumab treatment (Group A) compared with placebo (Group C)
Characterization of mean concentrations of anti-tetanus IgG during treatment with efalizumab compared with placebo, representing a secondary humoral immune response
Characterization of anti-pneumococcal antibody concentrations on FU Day 70 after pneumococcal vaccination on FU Day 42 compared with placebo
Percentage of subjects with positive skin test reactions to tetanus and Candida-recall antigens on FU Day 77 after washout from efalizumab compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dummer, M.D., Study Director — Genentech, Inc.